CLINICAL TRIAL: NCT00497250
Title: Phase I Study of Iressa and CRT/IMRT in Chinese Patients With IIIB/IV NSCLC After Failure of Platinum-Based Chemotherapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Guoliang Jiang, President of Cancer Hospital, Fudan University, Cancer Hospital, Fudan University, Shanghai, China
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDCA001
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Phase 1 Clinical Trials; Iressa; radiation therapy; Chinese; NSCLC; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Radiotherapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Thoracic RT for patients will start from 54Gy, and then escalate dose at 2Gy increment to 60Gy. At each dose level, 8 patients are required to complete RT without dose limiting toxicity(DLT). Evaluation will be done after 8 patients have completed the treatment.If there are >=2 DLT in the first 8 patients, the maximum tolerated dose (MTD) is achieved. If there is a single DLT revealed, an additional 8 patients will be recruited to that dose level. Should there be severe complication occurred again be at least 1 more DLT, then MTD is thought to be achieved.Hence,MTD will be achieved if at least 2 out of the first 8 patients have a DLT,or if a further 8 patents are recruited, >=2 out of 16 patients have a DLT. Concurrent with RT, patients will be given gefitinib 250 mg/day PO as well as same dose PO for 60 days after the completion of RT.
  Interventions: Drug: Gefitinib; Device: Radiation Therapy

INTERVENTIONS:
Drug: Gefitinib — gefitinib 250 mg/day,PO concurrent with RT and 250 mg/day,PO for 60 days after the completion of RT.
  Other Names: Iressa@
Device: Radiation Therapy — group 1.54Gy/27Fx concurrent with gefitinib group 2.56Gy/28Fx concurrent with gefitinib group 3.58Gy/29Fx concurrent with gefitinib group 4.60Gy/30Fx concurrent with gefitinib
  Other Names: 3-D CRT and IMRT

SUMMARY:
The primary objective of this study is to evaluate the tolerability and the maximum tolerated dose of Conformal or Intensity-Modulated Radiotherapy when given in combination with gefitinib 250mg in Chinese patients with IIIB or IV NSCLC after failure of platinum-based chemotherapy.

Secondary objectives of the study are to obtain the preliminary information on efficacy after concomitant treatment of gefitinib 250mg and radiotherapy in Chinese patients with IIIB or IV NSCLC after failure of platinum-based chemotherapy, as measured by RECIST criteria.

To determine the pattern of failure (e.g., local, regional, or distant metastasis) in patients treated with this regimen.

DETAILED DESCRIPTION:
Laboratory research has suggested that targeting specific signalling proteins would be well suited for selectively enhancing the tumor radiosensitivity. In human xenograft models (non-small cell lung cancer and breast cancer) treated with gefitinib and irradiation, combined therapy has shown a significant increase in tumor growth delay as compared with monotherapy of irradiation or gefitinib. The epidermal growth factor receptor tyrosine kinase inhibitor ZD1839 selectively potentiates radiation response of human tumors in nude mice, with a marked improvement in therapeutic index. The authors concluded that gefitinib profoundly enhanced the antitumor action of RT against the tested tumors without significant adverse effects, increasing the therapeutic selectively of ionizing radiation in certain model systems. Substantial benefits for this multimodality therapy in patients could be expected.

While there are no published data on the feasibility and efficacy of combined gefitinib and radiation therapy in Chinese population who might be susceptible to gefitinib monotherapy, clinical studies have demonstrated that combining gefitinib with external beam radiation to 66-74Gy and concurrent weekly chemotherapy after induction chemotherapy were tolerated without excessive toxicity. In the present trail, we hope to build on our own experience of using combined gefitinib and thoracic radiation with 3D-CRT or intensity-modulated radiotherapy (IMRT) technique in a phase I setting for stage IIIb and selected stage IV NSCLC. We will follow this treatment (RT and gefitinib) with 60 days gefitinib at standard systemic doses.

ELIGIBILITY:
Inclusion Criteria:

* Understand and willing to sign the consent
* Provision of study-specific written informed consent
* Chinese ethnicity
* Histological or cytological conformation of NSCLC(maybe from initial diagnosis of NSCLC or subsequent biopsy). Of note,sputum cytology alone is not acceptable. Cytological specimens obtained by brushing, washing and needle aspiration of a defined lesion are acceptable
* Stage IIIB or stage IV,excluding those with pericardial or uncontrolled (not stable in past 60 days) pleural effusion. Stage IV patients must either be symptomatic due to pulmonary malignancies or only have CNS or bone metastases if there is clinical evidence of stable disease (no steroid therapy or steroid dose being tapered) for ≥28 days.
* ≥ 1 prior chemotherapy regimen (at least one platinum-based) for treatment of their disease and will have been progressed or intolerant to their most recent prior chemotherapy
* FEV1≥ 1000cc (without bronchodilator)
* FEV1/FVC >0.7 (with or without bronchodilator) or post-bronchodilator FEV1/FVC ≤0.7 but FEV1≥ 50% of predicted value

  * 1 measurable lesion according to RECIST criteria
* Life expectancy of ≥24 weeks
* Zubord-ECOG criteria performance status0-2(Karnofsky>60%)
* Normal organ and marrow function as defined below:

  * Leukocytes≥3,000/µL
  * Haemoglobin≥9g/dL (prior to transfusions)
  * Absolute neutrophil count ≥1,500/µL
  * Platelets ≥100,000/µL
  * Total bilirubin<1.5 X upper limit of normal
  * AST (SGOT)/ALT (SGPT) ≤2.5 X institutional upper limit of normal
  * Creatinine ≤ 2.5 mg/dl.
* Recovery from any acute toxicity related to prior therapy(CTC<2)

Exclusion criteria:

* Prior iressa therapy or prior therapy with an experimental agent whose primary mechanism of action is inhibition of EGFR or Pan-HER family receptors or its associated tyrosine kinase
* Prior thoracic radiotherapy
* Prior palliative RT whose port involved the lung or mediastinum region
* Newly diagnosed CNS metastases that have not been treated with surgery and/or radiation
* Newly diagnosed painful bony metastases w/o cord compression yet not treated with surgery and/or radiation
* Evidence of visceral metastases
* <21 days since prior chemotherapy, immunotherapy, or biological systemic anticancer therapy
* <28 days since prior cranial and/or bone irradiation
* Unresolved chronic or late toxicity from previous anticancer therapy inappropriate for this study according to the investigator
* Allergic reactions attributed to compounds of similar chemical or biologic composition to iressa
* Other co-existing malignancies or malignancies diagnosed within the last 5 years except basal cell carcinoma or cervical cancer in situ
* Unable to ingest oral medications
* Any co-morbid pulmonary disease that may put the patient at risk of severe toxicities. Specially,

  * Clinically active interstitial lung disease unless due to uncomplicated progressive lymphangitic carcinomatosis (except chronic stable radiographic changes who are asymptomatic)
  * Severe chronic obstructive pulmonary disease (COPD) defined as post-bronchodilator FEV1/FVC ≤0.7 and FEV1 ≤ 50% of predicted value (American Thoracic Society (ATS) classification)
* Concomitant use of phenytoin, carbamazepine, rifampicin, barbiturates, or St.John's Wort
* Other uncontrolled intercurrent illness including, but not limited to, ongoing or active infection and psychiatric illness/social situations that would limit compliance with study requirements
* Surgical incision from major surgery not healed
* Bleeding after biopsy(except small biopsy)
* Use a non-approved or investigational drug within 30 days before Day 1 of the trial treatment
* No measurable disease
* Pregnancy or lactating
* Receiving other investigational agents or devices

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-03 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities per protocol | 3, 6 and 12 months

SECONDARY OUTCOMES:
Response rate, mortality | 3, 6 and 12 months
Pattern of failure(e.g., local, regional, or distant metastasis) | 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Jiang, MD, Principal Investigator — Fudan University Cancer Hospital, Department of Radiation Oncology; Min Fan, M.D., Principal Investigator — Fudan University Cancer Hospital, Department of Radiation Oncology; Xiaolong Fu, M.D, Principal Investigator — Fudan University Cancer Hospital, Department of Radiation Oncology
Locations (1):
- Fudan University, Cancer Hospital, Department of Radiation Oncology, Shanghai, China